CLINICAL TRIAL: NCT01167452
Title: Population Pharmacokinetic Analysis of Sulfamethoxazole and Trimethoprim in Normal Weight, Overweight, and Obese Volunteers
Brief Title: Effect of Weight and/or Obesity on Sulfamethoxazole and Trimethoprim Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ron Hall, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMA IRB A10-3592; 5UL1RR024982-02 (NIH)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Pharmacokinetics; MRSA; Tuberculosis; PCP
Keywords: Obesity; Pharmacokinetics; MRSA; Tuberculosis; PCP
MeSH Terms: conditions — Obesity; Tuberculosis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sulfamethoxazole/trimethoprim (Experimental): 2 DS tablets of sulfamehtoxazole/trimethoprim (1600 mg/320 mg)
  Interventions: Drug: Sulfamethoxazole/trimethoprim

INTERVENTIONS:
Drug: Sulfamethoxazole/trimethoprim — 2 DS tablets of trimethoprim/sulfamethoxazole x 1 dose

SUMMARY:
This study will find how weight affects the dosing of a drug called sulfamethoxazole and trimethoprim. Currently, the amount of sulfamethoxazole and trimethoprim a patient receives is the same regardless of the patient's weight. The entire cohort was analyzed for the study outcomes. BMI groups were for recruitment purposes only and were not used for ordinal data analysis.

All sulfamethoxazole and trimethoprim (Trade name is Bactrim or Septra) medication that you will receive in this study will be referred to as study medication within this informed consent form. This drug is a combination of two antibiotics, sulfamethoxazole and trimethoprim, which belongs to a class of medication known as "sulfones" and is approved by the US Food and Drug Administration (FDA) for the treatment of a wide variety of bacterial infections such as ear infections, urinary tract infections, bronchitis, traveler's diarrhea, and Pneumocystis carinii pneumonia. Sulfamethoxazole and trimethoprim is given orally.

DETAILED DESCRIPTION:
This study is designed to measure drug concentrations in the blood of volunteers administered a single oral dose of sulfamethoxazole and trimethoprim. The volunteers to be enrolled will not have ear infections, urinary tract infections, bronchitis, traveler's diarrhea, Pneumocystis carinii pneumonia, or any other bacterial infection. This is a single center study. A total of 36 adult volunteers will be consented for the study at the Clinical and Translational Research Center (CTRC). Volunteers will be recruited using IRB approved fliers. Volunteers will be admitted to the CTRC for an overnight stay. Half will be female and half male. Twelve volunteers will have a body mass index (BMI) less than 25 kg/m2, twelve will have a BMI 25-40 kg/m2, and twelve will have a BMI greater than 40 kg/m2. Volunteers will have height and weight measured after they have consented to participate. All volunteers will receive a single oral dose of sulfamethoxazole and trimethoprim of 1600 mg/320 mg. The volunteers will have blood drawn via an intravenous catheter just prior to the dose, and then at 1, 2, 4, 8, 12, and 24h after the drug dose. The intravenous catheter is then removed after the 24h blood draw, and the volunteer is discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age >18 years, of all racial and ethnic origins.
* We are recruiting 12 normal or underweight (BMI <25kg/m2), 12 overweight or obese (BMI 25-40 kg/m2), and 12 extremely obese (BMI > 40 kg/m2) for this study. This index is calculated using the volunteer's height and weight (Formula: weight (lb) / [height (in)]2 x 703). Half of each group will be male; the other half will be female.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of sulfamethoxazole and trimethoprim on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of sulfamethoxazole and trimethoprim, so that the pregnancy and post-partum state would be a confounding variable.
* Abnormal liver function tests: transaminases>10 times upper limit of normal, Alkaline phosphatase>5 times upper limit of normal, total bilirubin>5 times upper limit of normal.
* History of allergies to sulfones, sulfonamides or trimethoprim.
* Sulfones, sulfonamides or trimethoprim are contraindicated for any reason.
* Volunteers unwilling to comply with study procedures.
* Current suspected or documented ear infection, urinary tract infection, bronchitis, traveler's diarrhea, Pneumocystis carinii pneumonia, or any other bacterial infection.
* Volunteers with colon resection, gastric bypass, lap band, or any other conditions inhibiting gastric absorption of drug.
* Current or previous participation within 28 days of enrollment in another research study that involves the use of medication, contrast, or any other compound that may alter blood count and/or blood chemistry (liver function, kidney function or electrolyte balance), unless waved by PI.
* Donation of 450mL (one unit) of blood or more within 8 weeks (56 days) prior to study enrollment, unless waved by PI.
* Current use of medications contraindication with sulfamethoxazole/trimethoprim use: Bepridil, Cisapride, Dofetilide, Levomethadyl, Mesoridazine, Pimozide, Terfenadine, and Thioridazine. Other medications will be screened by study investigators to ensure the safety of research participants and maintain the quality of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hall, PharmD, MSCS, Principal Investigator — Texas Tech UHSC
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hall RG Nd, Pasipanodya JG, Meek C, Leff RD, Swancutt M, Gumbo T. Fractal Geometry-Based Decrease in Trimethoprim-Sulfamethoxazole Concentrations in Overweight and Obese People. CPT Pharmacometrics Syst Pharmacol. 2016 Dec;5(12):674-681. doi: 10.1002/psp4.12146. Epub 2016 Nov 21. PMID 27869362
- See also: Link to manuscript describing our findings — http://onlinelibrary.wiley.com/doi/10.1002/psp4.12146/full

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulfamethoxazole/Trimethoprim
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sulfamethoxazole/Trimethoprim: All volunteers received a single dose oral dose of TMP/SMX (1600 mg/320 mg).
Arm/Group | Sulfamethoxazole/Trimethoprim
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 34
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 37 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Elimination Rate Constants for Sulfamethoxazole and Trimethoprim
Time Frame: 24 hours
Measure: Median (Full Range); unit: hr-1
Groups:
- Sulfamethoxazole: Results from sulfamethoxazole analysis
- Trimethoprim: Results from trimethoprim analysis
Arm/Group | Sulfamethoxazole | Trimethoprim
Number analyzed (Participants) | 36 | 36
hr-1 | 0.060 [0.015 to 0.180] | 0.03 [0.02 to 0.14]
Statistical Analysis 1: Comparison: Sulfamethoxazole; We conducted a linear regression analysis of the log transformed elimination rate constant vs. the log transformed weight for each participant; Test type: Superiority or Other; p = 0.0004, Regression, Linear; Multivariate adaptive regression spline (MARS) analysis; Slope = -0.74, Standard Deviation 0.19
Statistical Analysis 2: Comparison: Trimethoprim; We conducted a linear regression analysis of the log transformed elimination rate constant vs. the log transformed body mass index for each participant; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Multiple Adaptive Regression Spline (MARS); Slope = -0.56, Standard Deviation 0.20

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Sulfamethoxazole/Trimethoprim: All volunteers received a single dose of TMP/SMX (1600 mg/320 mg).
Arm/Group | Sulfamethoxazole/Trimethoprim
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 4/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamethoxazole/Trimethoprim (N=36)
Headache (Nervous system disorders) | 3 (3) — Mild headache post-dose (possibly related) One person with a headache also had elevated blood pressure, skin irritation under the medical dressing over the IV line insertion site, and a mild rash (neck, ears); all deemed not related to study drug.
Fainting (Nervous system disorders) | 1 (1) — One person fainted during the screening blood draw, which we judged not to be related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No